CLINICAL TRIAL: NCT04056338
Title: Gut Microbiome and Gut Barrier Function in ICU Delirium Post Cardiac Surgery
Brief Title: Gut Microbiome and ICU Delirium Post Cardiac Surgeries
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018001113
Record Dates: First submitted 2019-07-31; First posted 2019-08-14 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Intensive Care Unit Delirium
Keywords: delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium: Patients with delirium as assessed by the bedside nurse using Confusion Assessment Method for the ICU.
- Non-delirium: Patients without delirium.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention.
  Groups: Non-delirium

SUMMARY:
ICU delirium are assessed by clinical nurses twice every day. Delirious patients are matched with patients according to their disease, gender and age range(±3 years). Stool samples for gene sequencing are collected. Gut barrier function are studied with several serum biomarkers (endotoxin, etc.). Ecological analyses, regression models and mediation equation will be performed.

DETAILED DESCRIPTION:
ICU delirium are assessed by clinical nurses twice every day using Confusion Assessment Method for the ICU (CAM-ICU). Delirious patients are matched with patients according to their disease, gender and age range(±3 years). Stool samples for gene sequencing are collected within 24 hours after surgeries. Gut barrier function are studied with several serum biomarkers (endotoxin, etc.). Ecological analyses, regression models and mediation equation will be performed.

ELIGIBILITY:
Inclusion Criteria:

* to have had heart valve surgery or coronary artery bypass grafting (CABG)
* to have no planned transfer to another ward or hospital within 24 hours after surgery
* to have no preoperative cognitive impairment and can speak and read Chinese
* more than 18 years old

Exclusion Criteria:

* to have a hearing or visual impairment that could impact delirium assessment
* to have a history of alcohol or drug abuse
* to have a preoperative intestinal irritation syndrome or history of gastrointestinal disease
* to have received antibiotics or probiotics within 28 days before admission
* to have a life expectancy less than 24 hours
* to have an experience of ICU hospitalization, mechanical ventilation in the past 30 days
* to have a cardiac surgery or hypoxic brain injury in the past 3 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac surgery and admitted to CSICU are recruited.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Gut microbiome | within 24 hours of delirium
  Rectal swabs or stool samples for bacterical DNA extraction and 16S rRNA gene sequencing will be collected. Diversity and composition of gut microbiome will be compared between delirious and non-delirious patients.

SECONDARY OUTCOMES:
Gut barrier biomarkers | within 24 hours of matched samples
  Blood sample will be collected to analyze the level of three gut barrier biomarkers (endotoxin, D-lactate and diamine oxidase).

CONTACTS AND LOCATIONS:
Overall Officials: Jingfen Jin, Study Director — SAHZU
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No